CLINICAL TRIAL: NCT00476385
Title: Usability and Acceptability of Stylomax® in Growth Hormone Deficient Children.
Brief Title: Practicability and Acceptability of Stylomax® in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8912
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- somatropine (Experimental)
  Interventions: Drug: somatropine

INTERVENTIONS:
Drug: somatropine — subcutaneous injections, 20 % less than the dosage of Maxomat 1.3 mg

SUMMARY:
Primary objective:

to evaluate the practicability and acceptability of STYLOMAX®, a new injection device for MAXOMAT®, in children, for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Children over 3 years of age with growth hormone deficiency, requiring treatment with MAXOMAT® according to the criteria of the MA.

Exclusion Criteria:

* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2003-06; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
practicability/acceptability of the Stylomax pen | at each visit

SECONDARY OUTCOMES:
tolerability : pain (evaluation on pain scale) | at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France